CLINICAL TRIAL: NCT00846833
Title: Phase I/II Study of Haploidentical Natural Killer Cell Infusion in Patients With Refractory or Relapsed Malignant Melanoma
Brief Title: Haploidentical NK Cell Infusion in Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Dae Seog Heo/Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0808-024-253
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma
Keywords: Melanoma, Experimental
MeSH Terms: conditions — Melanoma; Melanoma, Experimental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide, high-dose interleukin-2, NK cell (Experimental)
  Interventions: Biological: Haploidentical NK cell

INTERVENTIONS:
Biological: Haploidentical NK cell — 1. Collection of PBMCs by leukapheresis
  2. CD3+ depletion of apheresis product using CliniMACS®

SUMMARY:
We hypothesized that haploidentical NK cells kill tumor cells more efficiently than autologous NK cells, based on the missing-self hypothesis. Therefore, we performed this study to investigate the role of haploidentical NK cell therapy in patients with refractory or relapsed malignant melanoma.

DETAILED DESCRIPTION:
Human NK cells recognize and kill transformed cells in a MHC-unrestricted fashion, suggesting the role of cancer immunotherapy. However, autologous NK cells showed the lack of significant clinical effects, because they are inhibited by self MHC class I molecules, based on the missing-self hypothesis. Contrarily, haploidentical NK cells with KIR-ligand incompatibility can mediate graft-versus-leukemia effect and protect patients with acute myelogenous leukemia (AML) from graft-versus-host disease. In addition, adoptive transfer of haploidentical NK cells following high-intensity conditioning induced complete remission (26%) in poor-prognosis AML patients. Thus, this study was designed to investigate the role of adoptive NK cell therapy in patients with refractory or relapsed malignant melanoma using CD3+ depleting CliniMACS® system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or relapsed malignant melanoma
* Patients who received prior chemotherapy or immunotherapy
* Patients who have at least one haploidentical donor willing to donate
* ECOG performance status 0 or 1
* 18 - 75 years
* At least one measurable disease according to the RECIST criteria
* Patients with 45% or more left ventricular ejection fraction
* Patients with 50% or more predicted DLCO
* Adequate bone marrow function: absolute neutrophil count ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L; and hemoglobin ≥ 9 g/dL
* Adequate liver function: total bilirubin ≤ 1.0 x upper limit of the normal range (ULN); AST/ALT ≤ 2.5 x ULN; and alkaline phosphatase ≤ 2.5 x ULN
* Adequate renal function: serum creatinine ≤ 1.0 x ULN or creatinine clearance ≥ 60 mL/min/1.73m2
* At least 3 months of expected survival
* Patients who signed informed consent

Exclusion Criteria:

* Patients who received other chemotherapeutic agents within 30 days prior to study enrollment
* Patients who received adoptive cell therapy including hematopoietic stem cell transplantation
* Patients infected with HIV, HBV, or HCV
* Hypersensitivity to cyclophosphamide or interleukin-2
* Patients who received organ transplantation
* Patients who had arrhythmia or ischemic heart disease
* Pregnant or lactating women
* Patients with uncontrolled infection who did not respond to appropriate antimicrobial agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum-tolerated dose of haploidentical NK cells | 1 year

SECONDARY OUTCOMES:
To assess NK cell infusion-related toxicity | 2 years
To evaluate response rate | 2 years
To determine immune reconstitution after NK cell infusion | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dae Seog Heo, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea